CLINICAL TRIAL: NCT04078841
Title: Using ReaLife+ to Treat Post-Lyme Disease Syndrome
Brief Title: Treating Post-Lyme Disease Syndrome With Acetogenins
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Optimal Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RLP042019
Record Dates: First submitted 2019-08-31; First posted 2019-09-06 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Post-Lyme Disease Syndrome (PLDS)
MeSH Terms: conditions — Post-Lyme Disease Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ReaLife+ (RLP) (Active Comparator): Dietary Supplement: ReaLife+ (RLP) RLP is a dietary supplement containing Acetogenins, vitamin, mineral and amino acids
  Interventions: Dietary Supplement: ReaLife+ (RLP)
- Inert Brown Powder (Placebo Comparator): Brown powder
  Inert brown powder to look similar to RLP
  Interventions: Other: Inert Brown powder
- Control (No Intervention): Control

INTERVENTIONS:
Dietary Supplement: ReaLife+ (RLP) — RLP is a dietary supplement containing Acetogenins, vitamin, mineral and amino acids.
  Arms: ReaLife+ (RLP)
Other: Inert Brown powder — Brown powder Inert brown powder to look similar to RLP
  Arms: Inert Brown Powder

SUMMARY:
To access the effectiveness of Acetogenins in treating Post-Lyme Disease Syndrome (PLDS).

DETAILED DESCRIPTION:
To access the effectiveness of Acetogenins in treating Post-Lyme Disease Syndrome (PLDS). After failure of antibiotic therapy to relive persistent symptoms of Lyme Disease, the use of Acetogenins to elevate Post-Lyme Disease Syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. A positive Western Blot for Lyme Disease that has been treated with antibiotics but the symptoms persist post treatment.
2. Must be able to swallow and mixed powder drink.

   -

Exclusion Criteria:

1. Non Positive Western Blot test.
2. Positive Western Blot test where the indivual has not been treated with antibiotics.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Blood test | 3 months
  Western Blot showing "negative"
PROMIS Fatigue Scale | 3 months
  Self reported fatigue level changes as measured by the Patient-Reported Outcomes Measurement Information System, Fatigue Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Jeppsen, MD, Study Chair — IRB Chair
Locations (1):
- Optimal Health Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No